CLINICAL TRIAL: NCT06709807
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover Study to Evaluate the Food Effect on the Safety and the Pharmacokinetics of CKD-378 in Healthy Adult Volunteers
Brief Title: Clinical Study to Evaluate the Food Effect of CKD-378 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A129_04FDI2412
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fast-Fed (Experimental): Period 1: A single oral dose of 1 tablet under fasting condition, Period 2: A single oral dose of 1 tablet under fed condition
  Interventions: Drug: CKD-378 25/1000mg
- Fed-Fast (Experimental): Period 1: A single oral dose of 1 tablet under fed condition, Period 2: A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-378 25/1000mg

INTERVENTIONS:
Drug: CKD-378 25/1000mg — QD, PO

SUMMARY:
This study is a randomized, open-label, single dose, crossover study to evaluate the food effect of CKD-378 in healthy volunteers

DETAILED DESCRIPTION:
To 30 healthy subjects, following treatments are administered dosing in each period and wash-out period is 7 days.

Pharmacokinetic blood samples are collected up to 48hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who is 19 years of age or older at the time of the screening visit
2. Individuals who had 18.0 kg/m2 ≤ Body Mass Index(BMI) < 30.0 kg/m2 and total body weight ≥ 50 kg BMI = Weight(kg)/ Height(m)2
3. Individuals who do not have clinically meaningful congenital or chronic diseases and who do not have medical examination results (such as electroencephalogram, electrocardiogram, chest and gastroscopy or gastrointestinal radiography, if necessary) during screening visits
4. Individuals determined by investigators to be suitable for testing as a result of diagnostic tests and electrocardiogram tests, such as hematology tests, blood chemistry tests, serum tests, urine tests, etc
5. Individuals who agreed proper contraception during the study and did consent to not donation of sperm or eggs 7 days after the last dose of study drug
6. Individuals who signed an informed consent form after being fully informed of the study prior to participation, including the objective and content

Exclusion Criteria:

1. Individuals who has a history of gastrointestinal surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of drugs or has a gastrointestinal disease
2. Individuals who has used a drug metabolase-inducing and inhibiting drug such as barbitals within one month prior to the first dosing date or a drug that may interfere with this test within 10 days prior to the first administration of investigational product
3. Individuals who had been administered investigational product from other clinical study or bioequivalence study within the 6 months prior to the first administration of investigational product
4. Individuals who donated whole blood within the 8 weeks, or blood components within 2 weeks or had a blood transfusion within 4 weeks prior to the first administration of investigational product
5. Individuals who meets the following conditions within one month prior to the first administration of investigational product

   * Man: average alcohol consumption > 21 cups/weeks
   * Woman: average alcohol consumption > 14 cups/weeks
   * Smoking > 20 cigarettes
6. Patients with the following conditions

   * Patients with hypersensitivity to investigational product or biguanide drugs
   * Patients with acute or chronic metabolic acidosis including type 1 diabetes, lactic acidosis, comatose or not diabetic ketoacidosis, and patients with a history of ketoacidosis
   * Acute conditions that can affect renal functions such as moderate (stage3b) and severe renal impairment (glomerular filtration rate <45ml/min/1.73m2), dehydration, severe infection, cardiovascular despondency (shock), acute myocardial infarction, sepsis, etc
   * Patients with acute and unstable heart failure
   * Patients undergoing tests for intravenous administration of radioiodine contrast agents (e.g., intravenous urinary tract, intravenous cholangiography, angiography, computed tomography with contrast agents, etc.)
   * diabetic coma
   * Patients with severe infections or severe traumatic systemic disorders
   * Patients scheduled for surgery
   * Patients with malnutrition, starvation, weakness, pituitary dysfunction or adrenal insufficiency
   * Acute or chronic patients who can cause liver dysfunction, respiratory failure, and tissue hypoxia
7. Individuals with a clinically significant history of mental illness
8. Those who are deemed insufficient to participate in this clinical study by investigators
9. Pregnant women, women who may be pregnant, nursing women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-378 | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 24, 32, 48 hours
  Area under the CKD-378 concentration in blood-time curve from 0 to t
Cmax of CKD-378 | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 24, 32, 48 hours
  The maximum CKD-378 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Gwanak-gu, Seoul, South Korea